CLINICAL TRIAL: NCT02400060
Title: Increasing Adherence to Adjuvant Hormonal Therapy Among Breast Cancer Patients: Phase 2 - Pilot Test of Intervention for Feasibility
Brief Title: Telephone-Based Intervention in Increasing Adherence to Adjuvant Hormonal Therapy in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other)
Responsible Party: Principal Investigator, Michelle Naughton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-13252; NCI-2014-00809 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage 0 Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive (text messages and interactive exchanges) (Experimental): Patients receive daily text messages reminding them to take AHT and weekly interactive surveys delivered by a smart phone app for 3 months.
  Interventions: Behavioral: Telephone-Based Intervention; Other: Survey Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Behavioral: Telephone-Based Intervention — Receive text messaging
Other: Survey Administration — Ancillary studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot trial studies a telephone-based intervention to see if it increases adherence to adjuvant hormonal therapy in patients with breast cancer. Increasing communication between doctors and patients with breast cancer may help patients to better follow recommendations on taking adjuvant hormonal treatment medication. A telephone-based intervention may help to increase doctor-patient communication and patients' adherence to their prescribed medication.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Pilot test intervention effects on adherence to adjuvant hormonal therapy (AHT) and explore trends in the adherence outcomes by demographic and psychosocial factors defined as acceptance, continuation, and adherence.

SECONDARY OBJECTIVES:

I. Feasibility of study design defined as recruitment rate, rate of using intervention as instructed, rate of protocol completion, and completion of psycho-social questionnaires which have been associated with adherence to AHT in the existing literature (i.e., depression, social support, pain, stress, fatigue, quality of life, pill taking attitude and behavior, perceived risk of breast cancer recurrence).

TERTIARY OBJECTIVES:

I. Surveying patients and physicians regarding their comments on the intervention components (i.e., video, text messaging, and app [application]) and overall study participation.

OUTLINE:

Patients receive daily text messages reminding them to take AHT and weekly interactive surveys delivered by a smart phone app for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women are those who:

  * Are post-menopausal, verified by:

    * Post bilateral surgical oophorectomy; or
    * No spontaneous menses >= 1 year; or
    * No menses for < 1 year with follicle stimulating hormone (FSH) and estradiol levels in postmenopausal range, according to institutional standards
* Are diagnosed with primary breast cancer (BC) (stages I-III)
* Eligible to receive AHT (tamoxifen or an aromatase inhibitors [AI]) for the first time
* Completed all primary treatment
* Own a smartphone (in order to receive text messages and utilize the phone app)
* Agree to receive text messages on their smartphone over a 3-month period
* Provide consent and permission to review their medical records
* Plan to stay in the study area for 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Optimal usage of AHT (includes initiation, continuation and adherence) | Up to 3 months
  Descriptive statistics will be generated. Confidence intervals (95%) for the outcomes will be generated using the Clopper-Pearson method. Logistic regression will be used to explore whether any trends are observed in the outcomes by demographic or psychosocial factors. Mediation analyses will be conducted to determine if any of the psychosocial measures are mediators of compliance.
Acceptance assessed via medical records of receiving a prescription for AHT and filling it | Up to 3 months
  Descriptive statistics will be generated. Confidence intervals (95%) for the outcomes will be generated using the Clopper-Pearson method. Logistic regression will be used to explore whether any trends are observed in the outcomes by demographic or psychosocial factors. Mediation analyses will be conducted to determine if any of the psychosocial measures are mediators of compliance.
Continuation assessed via self-report of taking at least one dose per week | Up to 3 months
  Descriptive statistics will be generated. Confidence intervals (95%) for the outcomes will be generated using the Clopper-Pearson method. Logistic regression will be used to explore whether any trends are observed in the outcomes by demographic or psychosocial factors. Mediation analyses will be conducted to determine if any of the psychosocial measures are mediators of compliance.
Adherence assessed via self-report of taking the prescribed dose at least 6 of 7 days per week | Up to 3 months
  Descriptive statistics will be generated. Confidence intervals (95%) for the outcomes will be generated using the Clopper-Pearson method. Logistic regression will be used to explore whether any trends are observed in the outcomes by demographic or psychosocial factors. Mediation analyses will be conducted to determine if any of the psychosocial measures are mediators of compliance. Weekly compliance (number of days reported taking medication) via the text messaging system will be examined longitudinally to assess whether a change over time was observed.

SECONDARY OUTCOMES:
Change in biomarkers | Baseline to 3 months
  Comparisons (correlations, bivariate plots) will be made between the biomarkers and self-reported rates of usage to explore the feasibility of using a biomarker to measure optimal usage in future studies.
Patient and physician responses to the intervention and study participation | 3 months
  Descriptive statistics will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Naughton, PhD, MPH, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fletcher Allen Health Care-Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu